CLINICAL TRIAL: NCT00005478
Title: Precursors of CVD Risk Factors--Project Heartbeat
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4962; R03HL057101 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hypertension

SUMMARY:
To elucidate the changes in body size, composition, and configuration occurring in adolescence, because these are important precursors of change in blood pressure and blood lipids.

DETAILED DESCRIPTION:
BACKGROUND:

Project HeartBeat! was uniquely designed to investigate the course of change in cardiovascular disease risk factors and several categories of covariates, including the anthropometric indicators addressed in this study. The data pertained to the 678 participants who entered the Project in 1991-93 at ages 8, 11 or 14 years of age, of whom 49.1 percent were female and 20.1 percent were black. Of the 395 participants who became eligible for 10 or more 4-monthly examinations, 349 (88.4 percent) completed at least 10 occasions; 538 participants of 556 who were eligible for seven or more examinations (96.8 percent) completed at least seven. Multi-level (MLn) analytic methods previously tested with other data were utilized for this analysis.

DESIGN NARRATIVE:

Data from Project Heartbeat were analyzed. Hypotheses tested included: (1) the time patterns of change in several indicators of body size, composition and configuration over the period of observation; (2) the relations between the time patterns of change in these indicators and the corresponding patterns for change in selected endocrine factors; and (3) the explanatory contributions of energy intake and expenditure to variation between individuals in their observed time patterns of change in these indicators. The anthropometric indicators addressed were: weight (total mass), height, body mass index (BMI, wt/ht2), fat-free mass, fat mass, per cent body fat, and fat distribution (waist/hip ratio). Each of these indicators were examined first separately and then in relation to selected endocrinologic measures (testosterone, estradiol, and DHEAS) and to energy intake and expenditure (from interview histories of diet and physical activity). Existing data from up to twelve 4-monthly examinations over the age range from 8-17 years conducted in Project HeartBeat! were analyzed.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1996-09; Study Completion 1998-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darwin Labarthe — University of Texas